CLINICAL TRIAL: NCT03721822
Title: Measurement of Pulmonary Inflammation Using 18F-NOS Positron Emission Tomography (PET/CT) in E-cigarette Users
Brief Title: Imaging Sex Differences in Smoking-Induced Pulmonary Inflammation
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 831205
Record Dates: First submitted 2018-10-25; First posted 2018-10-26 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Smoking, Cigarette; Smoking E-cigarette; Healthy Volunteer
MeSH Terms: conditions — Cigarette Smoking | interventions — Fluorine-18

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Traditional Cigarette Smokers (Experimental): Reported current cigarette smoking of at least 5 cigarettes per day, 5 days per week for the past 1 year with no history of e-cigarette use (cannabis or nicotine) during the 30 days prior to study enrollment
  Interventions: Drug: [18F]NOS
- Non-Smokers (Experimental): Reported non-smoking history or < 100 lifetime cigarettes, < 100 e-cigarette use episodes and < 100 lifetime cannabis use episodes
  Interventions: Drug: [18F]NOS
- Nicotine Vapers (Experimental): Reported current e-cigarette use of nicotine at least 5 days per week for the past year with no current combustible cigarette use, cannabis vaping or cannabis smoking during the 30 days prior to study enrollment
  Interventions: Drug: [18F]NOS
- Cannabis Vapers (Experimental): Reported current e-cigarette use of cannabis at least 5 days per week for the past year, no current combustible cigarette use, cannabis smoking or nicotine vaping during the 30 days prior to study enrollment
  Interventions: Drug: [18F]NOS
- Dual Smokers/Vapers (Experimental): Reported current e-cigarette use of cannabis and/or nicotine at least 5 days per week for the past year with cigarette or cannabis smoking during the 30 days prior to study enrollment
  Interventions: Drug: [18F]NOS
- Poly-use nicotine and cannabis group (Experimental): Poly-use nicotine and cannabis group: current e-cigarette use of nicotine and/or cigarette use (5 cigarettes per day) and/or use of cannabis, at least 4 days per week during the 30 days prior to study enrollment.
  Interventions: Drug: [18F]NOS

INTERVENTIONS:
Drug: [18F]NOS — [18F]NOS is an investigational radiotracer which each subject will have one [18F]NOS positron emission tomography/computed tomography (PET/CT) scan performed.
  Other Names: [18F]-6-(2-fluoro-propyl)-4-methylpyridin-2-amine

SUMMARY:
The purpose of this research is to measure the extent of lung inflammation between different groups of participants using a radioactive tracer called [18F]NOS. A radioactive tracer is a type of imaging drug that is labeled with a radioactive tag and injected into the body.

DETAILED DESCRIPTION:
This study will see how the tracer is taken up in the lungs using an imaging scan called Positron Emission Tomography / Computed Tomography (PET/CT). [18F]NOS is an experimental radioactive molecule used in PET imaging to measure inflammation in various organs in the body. Investigators are interested in studying whether there are differences in lung inflammation between E-cigarette users (vapers) cigarette smokers and non-smokers. [18F]NOS has not yet been approved by the Food and Drug Administration (FDA) for use except in a research study. The use of [18F]NOS in this study is allowed under an Investigational New Drug Application approved by the FDA.

Investigators are also going to be studying how the information from the PET/CT scan compares to other markers of inflammation in the blood. During the PET scan, Investigators will image Brain and Lungs in order to see if there is a difference between inflammation seen in the brain and the lungs and if these differences change depending on whether a subject is a smoker, e-cigarette user or non-smoker.

Consented participant in this study will undergo one (1) experimental [18F]NOS PET/CT scan. During the scan, PET/CT images will be taken of participant chest/torso in order to capture their lungs and a short image will be taken of their brain. Blood samples will be taken at various time points to test for markers of inflammation and to measure the concentration of the tracer in participants blood during the scan and participants will undergo some specific psychological questionnaires and tasks.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be 18-45 years of age
2. Subject must meet one of the following criteria:

   NIC vapers: current e-cigarette use of nicotine at least 5 days per week for the past year, no current combustible cigarette use, cannabis vaping, or cannabis smoking during the 30 days prior to study enrollment

   CAN vapers: current e-cigarette use of cannabis at least 5 days per week for the past year, no current combustible cigarette use, cannabis smoking, or nicotine vaping during the 30 days prior to study enrollment

   Cigarette smokers: current cigarette smoking of at least 5 cigarettes per day, 4 days per week for the past year with no e-cigarette use (cannabis or nicotine) during the 30 days prior to study enrollment

   Dual combustible and e-cigarette users: current e-cigarette use of cannabis and/or nicotine at least 5 days per week for the past year with cigarette or cannabis smoking during the 30 day prior to study enrollment

   Non-Smokers: reported non-smoking history or < 100 lifetime cigarettes, < 100 e-cigarette use episodes, and < 100 lifetime cannabis use episodes
3. Participants must be informed of the investigational nature of this study and be willing to provide written informed consent and participate in this study in accordance with institutional and federal guidelines prior to study-specific procedures.

Exclusion Criteria:

1. Females who are pregnant or breast feeding at the time of screening will not be eligible for this study; a urine pregnancy test will be performed in women of child-bearing potential at screening and on scan day.
2. Current untreated and unstable diagnosis of substance use disorder, except nicotine use disorder or cannabis use disorder
3. Positive urine drug screen for opiates, methamphetamine or cocaine at screening
4. Current unstable and/or untreated major depression or psychotic disorder per medical record review or self-reported
5. Use of inhaled or oral corticosteroids or anti-inflammatory medications per medical record review or self-report
6. History of lung trauma
7. Active (or within the previous 4 weeks of screening) lung infection or lung disease that impact uptake of [18F]NOS (e.g. tuberculosis, cystic fibrosis)
8. Inability to tolerate imaging procedures in the opinion of an investigator or treating physician
9. Any current or past medical condition, illness, or disorder as assessed by medical record review and/or self-reported that is considered by a physician investigator to be a condition that could compromise participant safety or successful participation in the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-10-23 (Actual); Primary Completion 2026-10-23 (Estimated); Study Completion 2026-10-23 (Estimated)

PRIMARY OUTCOMES:
lung inflammation using [18F]NOS PET/CT | 3 years
  lung inflammation using [18F]NOS PET/CT and compare uptake in ENDS users to traditional cigarette smokers and non-smokers.

SECONDARY OUTCOMES:
relationship between [18F]NOS uptake and peripheral inflammatory biomarkers | 3 years
  relationship between [18F]NOS uptake measures and established peripheral inflammatory biomarkers (e.g. C-reactive protein and Il-6).
differences in brain inflammation between three cohort using [18F]NOS PET/CT] | 3 years
  Using [18F]NOS PET/CT to explore relative differences in brain inflammation between ENDS users, traditional cigarette smokers and non-smokers.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Dubroff, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States